CLINICAL TRIAL: NCT07135531
Title: Continuous Glucose Monitoring in an Underserved Population: Impact on Glucose Control, Patient Reported Outcomes, Healthcare Utilization, and Long Term Complications
Brief Title: Continuous Glucose Monitoring (CGM) in an Underserved Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2024-1872
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Diabetes; Diabetes Mellitus; Diabetes Type 2
Keywords: Medicaid; Underinsured; Continuous glucose monitoring; Uninsured
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Self-Monitoring of Blood Glucose (SMBG) (Placebo Comparator): The study participants will be randomized to the self-monitoring group (control) after a period of two-week run-in and followed for 6 months. They will be given an opportunity to wear the CGM sensor for 3 months at the conclusion of the 6-month follow-up as an optional follow-up.
  Interventions: Device: Continuous Glucose Monitoring (CGM)
- Continuous Glucose Monitoring (CGM) (Active Comparator): The study participants will be randomized to the continuous glucose monitoring group (intervention).
  Interventions: Device: Continuous Glucose Monitoring (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitoring (CGM) — Continuous glucose monitors will be placed subcutaneously every 14 days.

SUMMARY:
The investigators aim is to conduct a randomized clinical trial in an underserved population who are either uninsured or on Medicaid and taking at least one injection of insulin daily. The investigators believe that this study will lead to considerable alleviation of health disparities and provide better care for an underserved population. This will be a pilot study to evaluate the feasibility of such a trial in this population before doing a larger multicenter trial.

DETAILED DESCRIPTION:
This study is a randomized open label trial with study participants being randomized to either a continuous glucose monitoring group (intervention) or a self-monitoring group (control) after a period of two-week run-in and followed for 6 months. All participants regardless of assignment will be provided diabetes education. Participants randomized to the self-monitoring group will be given an opportunity to wear the CGM sensor for 3 months at the conclusion of the 6-month follow-up as an optional follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Type 2 diabetes mellitus
* HbA1C ≥ 7.5%
* At least on 1 insulin injection therapy daily
* Patients established with primary care clinic or endocrinology clinic or diabetes clinics in the New Orleans and surrounding areas
* Patients with Medicaid or free care or uninsured
* Patients must be able to speak and understand English and be capable of providing informed consent to participate in the study

Exclusion Criteria:

* Type 1 diabetes mellitus
* Currently on CGM or using insulin pump
* Advanced renal disease or Estimated Glomerular Filtration Rate (eGFR) <40
* Serious co-morbidities which in the investigator's opinion, will make it challenging for patients to participate
* The patient has been diagnosed with end-stage renal disease, is on dialysis, or has had a kidney transplant, Hemoglobinopathies, iron therapy or other condition that interferes with HbA1c measurement
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated hemoglobin (HbA1c) between baseline and 6-month visits for both groups | Baseline, 6 months
  The investigators will take blood samples at baseline and at the 6 months visit to measure the HbA1c levels. Change in the level of HbA1c at 6 months will be compared between the 2 groups to assess the outcome.

SECONDARY OUTCOMES:
Change in Time in Range (TIR) | Baseline, 6 months
  TIR is a percentage of time that a person with diabetes spends within their target blood glucose range. The investigators will review the data from the CGM devices and assess if there are any changes in the TIR between the 2 groups at baseline and at 6 months. The higher the percentage is for TIR, the better the blood glucose control is for patients.
Change in documented hypoglycemia <70 mg/ dl and severe hypoglycemia - <54 mg/dl | Baseline, 6 months
  The investigators will measure the change in documented hypoglycemia and severe hypoglycemia in patients in both groups at baseline and at 6 months. The lower the numbers of the hypoglycemia incidences, the better the outcome is.
  Documented hypoglycemia and severe hypoglycemia will be measured as a percentage of time that a person with diabetes below their target blood glucose range.

CONTACTS AND LOCATIONS:
Overall Officials: Shaveta Gupta, MD, Principal Investigator — Tulane University
Locations (1):
- University Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No